CLINICAL TRIAL: NCT05035238
Title: Evaluation of the Efficacy, Safety and Immunogenicity of Inactivated COVID 19 Vaccine (TURKOVAC Inactive) in Healthy Population of 18 and 64 Years of Age (Both Inclusive): a Randomized, Double-blind, Phase IIb Clinical Trial
Brief Title: Evaluation of the Efficacy, Safety and Immunogenicity of Inactivated COVID 19 Vaccine(TURKOVAC) in Healthy Population of 18 and 64 Years of Age (Both Inclusive):a Randomized, Double-blind, Phase IIb Clinical Trial
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: the clinical trial did not initiated
Sponsor: Health Institutes of Turkey (Other Government)
Collaborators: Mene Research (Other); TC Erciyes University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TSB-VAC-COV-TUR-KF2B.03
Record Dates: First submitted 2021-09-01; First posted 2021-09-05 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2021-09

CONDITIONS: Covid19
Keywords: Inactivated vaccine; Phase IIb; Severe acute respiratory syndrome
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Intervention Model Description: Each subject will receive triple intramuscular dose of TURKOVAC 3 µg/0.5 mL or 4,5 µg/0.5 mL Vaccine on Day 0, Day 28, and Day 120. 200 healthy subjects in both genders will be dosed in double blinded groups with 1:1 randomization ratio.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Active Comparator): 3 μg / 0.5 mL
  Interventions: Biological: Triple dose vaccination by inactivated Covid19 vaccine
- Arm 2 (Active Comparator): 4,5 μg / 0.5 mL
  Interventions: Biological: Triple dose vaccination by inactivated Covid19 vaccine

INTERVENTIONS:
Biological: Triple dose vaccination by inactivated Covid19 vaccine — triple dose intramuscular vaccine on Day 0, Day 28, and Day 120.

SUMMARY:
The objective of this study is to evaluate the efficacy, immunogenicity and safety of two different strengths (3 µg/0.5 mL and 4,5 µg/0.5 mL) of inactivated COVID 19 Vaccine- TURKOVAC in healthy subjects following 3rd vaccination to demonstrate clinical evidence in prophylaxis of COVID 19.

DETAILED DESCRIPTION:
This is a double-blind, triple dose, parallel, randomized design study comparing two different dose levels and immunization regimen of a novel COVID-19 vaccine candidate - TURKOVAC - against SARS-CoV-2 infection, to assess the efficacy and safety of these vaccine strengths after 3rd dose vaccination. This study will also provide more data to assess the efficacy of the 3rd dose vaccination (booster dose) for COVID-19 prophylaxis including comparison to a cohort of standard convalescent serum samples obtained from World Health Organization (WHO).

This study will be completed in 12 months.

ELIGIBILITY:
Inclusion criteria:

1. Caucasian race, 18 to 64 years of age male or female (both inclusive),
2. accepting not to participate in another COVID-19 vaccine study until the end of the study,
3. voluntarily gives written informed consent prior to any study-related procedures.
4. has a Body Mass Index (BMI) of 18.5-32.0 kg/m2-both inclusive,
5. has a normal/acceptable ECG result
6. for female volunteers of childbearing potential, a negative serum pregnancy test within seven days before vaccination:

   * Females of childbearing potential are defined as fertile following menarche and until becoming postmenopausal or permanently sterile. (Postmenopausal is defined as absence of vaginal bleeding or spotting for at least one year. Permanently sterile is defined as having had a hysterectomy, bilateral salpingectomy, or bilateral oophorectomy.)
7. for female volunteers of childbearing potential, volunteers who do not plan to get a child in the next one year; a willingness to use highly effective* contraceptive measures adequate to prevent a new pregnancy for the duration of the study, including for at least 12 months after receiving the first dose of study vaccination. For women with reproductive potential who use a hormonal method of contraception, concurrent use of a second (barrier) method is recommended.

   * Highly effective methods of birth control are defined as those that result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly (e.g. implants, injectables, oral contraceptives, some intrauterine devices, bilateral tubal occlusion, true sexual abstinence in line with the preferred and usual lifestyle of the volunteer, or vasectomized partner).
8. for sexually active males, a willingness to use contraceptive measures, e.g. a condom, for the duration of the study, including for at least three months after receiving the last dose of study vaccination. In addition, males must agree not to donate sperm over the same study period and for at least three months after receiving the last dose of study vaccination.
9. anti-SARS CoV 2 total antibody (including COVID-19 IgG and/or IgM) negative in serum.
10. physical examination, if indicated only (general state and abnormal findings per system: endocrine/metabolic, allergies, drug sensitivities, head, neck, eyes, ears, nose, throat, cardiovascular, respiratory, gastrointestinal, hepatic/biliary, urogenital, musculoskeletal, lymph nodes, skin, and neurological/psychiatric) should be normal/acceptable.

Exclusion criteria:

1. clinically significant infection or other acute illness not due to SARS-CoV-2, including fever ≥ 37.4°C within 24 hours prior to the planned study vaccination.
2. had close contact to persons with confirmed SARS-CoV-2 infection within 14 days prior to screening Visit 1.
3. has participated in a clinical study involving an investigational SARS-CoV-2 vaccine.
4. has a history of SARS-CoV-1 or MERS infection (self-reported).
5. positive test results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
6. has received any vaccine within 30 days prior Visit 1 other than the study intervention, with the exception of the seasonal influenza vaccination.
7. has abnormal findings in any required study investigations (including medical history, vital signs, physical examination, and clinical laboratory) considered clinically relevant by the Investigator.
8. with either medical history of or present acute or progressive, unstable or uncontrolled clinical conditions that pose a risk for participation or completion of the study, based on Investigator's clinical judgement.
9. with underlying diseases with a high risk of developing severe COVID-19 symptoms if infected.
10. has a history of malignancy in the past five years other than squamous cell or basal cell skin cancer. If there has been surgical excision or treatment more than five years ago that is considered to have achieved a cure, the subject may be enrolled. A history of hematologic malignancy is a permanent exclusion. Subjects with a history of skin cancer must not be vaccinated at the previous tumor site.
11. has a known or suspected defect of the immune system, such as subjects with congenital or acquired immune deficiency.
12. received immuno-suppressive therapy within four weeks prior to Visit 1 or receipt of immunosuppressive therapy is expected during the study.
13. has a history of any vaccine related contraindicating event.
14. presents with clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
15. has donated blood, blood fractions or plasma within four weeks prior to Visit 1 or received blood-derived products (e.g., plasma) within 12 weeks prior to Visit 1 in this study or plans to donate blood or use blood products during the study.
16. with clinically significant bleeding disorder (e.g., factor deficiency, coagulopathy or platelet disorder) or prior history of significant bleeding or bruising following IM injections or venipuncture.
17. has a rash, dermatological condition or tattoos that would, in the opinion of the Investigator, interfere with injection site reaction rating.
18. has a known or suspected problem with alcohol, caffeine or drug abuse as determined by the Investigator.
19. has any condition that, in the opinion of the Investigator, may compromise the subject's well-being, might interfere with evaluation of study endpoints, or would limit the subject's ability to complete the study.
20. has participated in another clinical study involving an investigational medicinal product (IMP) or device within 4 weeks prior to Visit 1 or is scheduled to participate in another clinical study involving an IMP, or device during this study.
21. blood pressure, after resting for five min, higher than 140/90 or lower than 100/60 mm Hg.
22. pulse rate outside the range of 50 - 100 beats/min OR respiratory rate outside the range of 15 - 18 breathings /min, after resting for five min.
23. laboratory values (blood/serum examination: sodium, potassium, calcium, total protein, albumin, glucose, creatinine, BUN, total bilirubin, AST, ALT, GGT, ALP, hemoglobin, hematocrit, erythrocytes, leukocytes, platelet count; HBsAg, HIV-Ab, HCV-Ab, urinalysis if requested) outside normal range with clinical relevance at entry.
24. intake or administration of OTC medication (including herbal remedies) which may have an effect on the study according to the investigator within 2 weeks prior to the start of the study.
25. legal incapacity and/or other circumstances rendering the subject unable to understand the nature, scope and possible consequences of the study.
26. is a member of the team conducting the study or in a dependent relationship with one of the study team members.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy Outcome | on day 14 and 28 after 3rd vaccination
  comparison of the seroconversion rate-at least 4-fold rise of antibody concentration/titre from pre- to post-vaccination
Efficacy Outcome | on day 14 and 28 after 3rd vaccination
  comparison of antibody concentrations (GMC) or titres (GMT) from pre- to post-vaccination; Specific ELISA antibody titres against SARS-COV-2 spike glycoprotein
Efficacy Outcome | on day 14 and 28 after 3rd vaccination
  comparison of neutralizing antibodies and cytokine (TNF-alpha, IFN-γ, IL-2, IL-4, IL-5 and IL-6) from pre- to post-vaccination
Efficacy outcome | on day 14 and 28 after 3rd vaccination
  • comparison of antibody responses levels of minimum of 40 participants to convalescent serum plasma obtained from WHO from pre- to post-vaccination

SECONDARY OUTCOMES:
Safety outcome | 12 months
  Adverse events and safety laboratory results

CONTACTS AND LOCATIONS:
Overall Officials: ZAFER SEZER, Principal Investigator — Erciyes University Hakan Çetinsaya Iyi Klinik Uygulama ve Arastirma Merkezi, IKUM (Center for GCP)
Locations (1):
- Erciyes University Hakan Çetinsaya Iyi Klinik Uygulama ve Arastirma Merkezi, IKUM (Center for GCP), Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No